CLINICAL TRIAL: NCT06306482
Title: Restriktif ve Obstrüktif Akciğer Hastalıklarında Postür ve Postürle İlişkili Faktörlerin Belirlenmesi
Brief Title: Determination of Posture in Patients With Restrictive and Obstructive Lung Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, Principal investigator; PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: SBA 23/390
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Lung Diseases, Obstructive; Lung Diseases; Postural; Defect
MeSH Terms: conditions — Lung Diseases, Obstructive; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Patients with chronic obstructive lung disease, asthma, cystic fibrosis and bronchiectasis.
- Group B: Patients with diffuse parenchymal lung diseases
- control group: healthy aged matched individuals.

SUMMARY:
The aim of this study is to determine posture and posture related factors in patients with restrictive and obstructive lung disease.

DETAILED DESCRIPTION:
It is aimed at investigating posture and posture related factors according to both type of disease and severity of disease in patients with restrictive and obstructive lung disease. The secondary purpose is to develop a model that determines correlations between posture and functional exercise capacity, respiratory and peripheral muscle strength, tightness of muscle, balance, and physical activity for each disease that will be included in this study. In accordance with these purposes, for each group, at least 15 patients with obstructive and restrictive lung disease will be included according to the inclusion and exclusion criteria for each disease, and 15 healthy controls will be included. Tests and questionnaires will be used in order to determine the severity of diseases. Lung function test and respiratory and peripheral muscle strength test will be performed. Time and Go test (TUG) and One minute sit to stand test will be performed. To evaluate the accessory respiratory muscles, a muscle tightness test will be performed for each muscle. Six Minute Walk Test (6 MWT) will be performed with an armband that measures energy expenditure for functional exercise capacity. To evaluate posture, the Corbin Postural Assessment Scale and photographic analysis will be used. Photographical analysis using software in lateral, posterior, and anterior views will be used for the cervical, thoracic, and lumbar regions. For angular and length measurements, anatomical landmarks will be determined and calculated in the regions. According to the results to be obtained, changes in posture according to the regions and posture related factors will be determined for each disease. It will guide professional working in this field.

ELIGIBILITY:
Inclusion Criteria:

Chronic Obstructive Pulmonary Disease Group Inclusion Criteria:

* Over 55 years old,
* Stage 1-2-3-4 according to the GOLD,
* Being clinically stable for the last 4 weeks.

Chronic Obstructive Pulmonary Disease Group Exclusion Criteria:

* Receiving long-term oxygen therapy,
* Having central and peripheral vestibular disease,
* Communication problems, known mental and cognitive problems,
* Having undergone any surgical intervention related to the spine within the last six months,

Inclusion Criteria for the Cystic Fibrosis Group:

* Being diagnosed with CF as a result of two sweat tests,
* Being over 18 years old.

Cystic Fibrosis Group Exclusion Criteria:

* Being in acute pulmonary exacerbation period,
* Receiving long-term oxygen therapy,
* Having undergone any surgical intervention related to the spine within the last six months,

Inclusion Criteria for the Asthma Group:

* Diagnosed with asthma according to the Global Strategy for the Prevention and Treatment of Asthma (GINA),
* Clinically stable for the last 1 month
* Being over 18 years old.

Asthma Group Exclusion Criteria:

* Change in medication for the last 1 month.
* Having undergone any surgical intervention related to the spine in the last six months,

Inclusion Criteria for Bronchiectasis Group:

* Being over 18 years old,
* Being diagnosed with bronchiectasis other than cystic fibrosis,
* Being clinically stable for the last 1 month.

Bronchiectasis Group Exclusion Criteria:

* Receiving long-term oxygen therapy,
* Having undergone any surgical intervention related to the spine in the last six months.

Diffuse Parenchymal Lung Diseases Inclusion Criteria:

* Being diagnosed with diffuse parenchymal lung according to American Thoracic Society/European Respiratory Society (ATS/ERS) criteria,
* Being over 18 years old,
* Having volunteered to participate in the research,
* To be clinically stable and to have comorbid conditions (such as hypertension, diabetes) under control,

Diffuse Parenchymal Lung Diseases Exclusion Criteria:

* Having undergone any surgical intervention related to the spine within the last six months,
* Having exacerbation in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obstructive and restrictive lung disease and healthy controls will be included in this study according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-03-07 (Estimated); Primary Completion 2025-03-07 (Estimated); Study Completion 2026-03-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of horizontal alignment of the head anterior view | 1 day
  Angle between left and right tragus and horizontal will be measured via photographic analysis
Evaluation of horizontal alignment of the trunk anterior view | 1 day
  Angle between left and right acromion and horizontal will be measured via photographic analysis Angle between left and right anterior superior iliac spine and horizontal will be measured via photographic analysis.
  Angle between left and right acromion and left and right anterior superior iliac spine will be measured via photographic analysis.
Evaluation of horizontal alignment of the head lateral view | 1 day
  Angle between left-right tragus and C7 spinous process and horizontal will be measured via photographic analysis.
Evaluation of vertical alignment of the head lateral view | 1 day
  Angle of acromion and tragus (left-right) and vertical will be measured via photographic analysis.
Evaluation of horizontal alignment of the trunk lateral view | 1 day
  Angle between anterior superior iliac spine and posterior superior iliac spina and horizontal will be measured via photographic analysis.
Evaluation of vertical alignment of the trunk lateral view | 1 day
  Angle between acromion and greater trochanter and vertical will be measured via photographic analysis.
Evaluation of horizontal asymmetry trunk in posterior view | 1 day
  Horizontal asymmetry of scapula in relation to T3 spinous process will be measured via photographic analysis.
Evaluation of scapulae | 1 day
  Investigation of posture by photographic analysis upward rotation/ anterior tilt/internal rotation of scapula, scapular elevation, and scapular abduction evaluations will be measured photographic analysis.
Posture | 1 day
  Posture will be examined via the Corbin Postural Assessment Scale. The total points of the Corbin Postural Assessment Scale range from 0 to 28 points. A higher point represents worse posture.

SECONDARY OUTCOMES:
Functional exercise capacity | 1 day
  Functional exercise capacity will be determined via Six Minute Walk Test.
Respiratory Muscle Strength | 1 day
  Respiratory muscle strength will be assessed using a mouth pressure device according to American Thoracic Society/ European Respiratory Society guidelines.
Lung function | 1 day
  Lung function will be assessed via a spirometer according to American Thoracic Society/ European Respiratory Society guidelines.
Dyspnea | 1 day
  Dyspnea will be assessed via The Modified Medical Research Council. The Modified Medical Research Council consists of five grades. A higher grades represents severe dyspnea level.
Peripheral muscle strength | 1 day
  Peripheral muscle strength will be assessed via hand dynamometer.
Lower extremity capacity | 1 day
  One minute sit to stand test will be used for lower extremity capacity.
Energy expenditure | 1 day
  An armband will be used to assess energy expenditure during six minute walk test.
Balance and Fall risk | 1 day
  Time up and go test will be used to assess balance and fall risk
Tightness of muscle | 1 day
  Pectoralis minör, pectoralis majör, adductor and internal rotator muscles, sternocleidomastoideus, and trapezius muscle tightness tests will be performed during musculoskeletal examination using a tape.
Severity of disease for patients with COPD | 1 day
  Global Initiative for Chronic Obstructive Pulmonary Disease, Global Initiative for Chronic Obstructive Pulmonary A,B,E assessment Tool will be used for patients with COPD. According to the Global Initiative for Chronic Obstructive Pulmonary Disease, the severity of airflow limitation (Forced Expiratory Volume in 1 s) was determined as mild (≥ 80%), moderate (50-80%), severe (30-50%), and very severe (<30%). According to Global Initiative for Chronic Obstructive Pulmonary ABE assessment Tool, patients classified group A, B, and E using symptom status and airflow limitation.
Severity of disease for patients with bronchiectasis | 1 day
  Patients with non- cystic fibrosis bronchiectasis will be classified into three groups according to the Forced Expiratory Volume in 1 s, Age, Chronic colonisation, Extension, Dyspnea level. According to this classification system, patients will be classified as 0-2 points mild, 3-4 moderate, 5-7 severe bronchiectasis.
Diffusion capacity for patients with diffuse parenchymal lung diseases | 1 day
  Carbon Monoxide Diffusion Capacity test with single breath method will be used for patients with diffuse parenchymal lung diseases.
Symptoms for patients with COPD | 1 day
  Chronic Obstructive Pulmonary Disease Assessment Test will be used to determined symptoms in patients with COPD. The total score of Chronic Obstructive Pulmonary Disease Assessment Test changes from 0 to 40 points, and 10 points is the accepted cut-off point for COPD.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Aynur Demirel, Ankara
  - Hacettepe University, Ankara